CLINICAL TRIAL: NCT01563302
Title: A Phase 1/2 Study of ISIS 481464, an Antisense Oligonucleotide Inhibitor of STAT3, Administered to Patients With Advanced Cancers
Brief Title: Phase 1/2, Open-label, Dose-escalation Study of IONIS-STAT3Rx, Administered to Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISIS 481464-CS1
Record Dates: First submitted 2012-02-13; First posted 2012-03-26 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Advanced Cancers; DLBCL; Lymphoma
Keywords: Advanced Cancers; DLBCL; Advanced Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): IONIS-STAT3Rx
  Interventions: Drug: IONIS-STAT3Rx

INTERVENTIONS:
Drug: IONIS-STAT3Rx — Three-hour IV infusions on Cycle 0 Days 1, 3, 5, and weekly three-hour IV infusions in Cycles 1 and beyond, on Days 1, 8, and 15 of each cycle.
  Other Names: ISIS 481464

SUMMARY:
This is a Phase 1/2, open-label, dose-escalation, dose-expansion study for the treatment of patients with advanced cancers. Eligible patients with DLBCL or other advanced lymphomas will be enrolled into the dose-expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Tumors that are relapsed or refractory to at least 1 prior anti-cancer systemic therapy and for which no standard therapy exists
* Expansion cohort only: Advanced lymphoma confirmed by histopathology
* Measurable or evaluable disease according to RECIST for solid tumors or according to IWRC for NHL tumors
* ECOG Performance Status less than or equal to 2
* Life expectancy greater than 12 weeks in the opinion of the Investigator

Exclusion Criteria:

* Any active or uncontrolled infection
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months prior to screening
* Prior radiation therapy, chemotherapy, hormonal therapy, or immunotherapy within 4 weeks prior to screening or 5 half-lives of the therapy, whichever is shorter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2016-03-23 (Actual); Study Completion 2016-03-23 (Actual)

PRIMARY OUTCOMES:
Safety of IONIS-STAT3Rx in patients with Advanced Cancers | Approximately 28 days after last dose of IONIS -STAT3Rx
Maximum-tolerated dose (MTD) of IONIS-STAT3Rx in patients with Advanced Cancers. | Approximately 28 Days
  Highest dose level at which no more than 1 out of 6 patients develops a DLT

SECONDARY OUTCOMES:
Clinical activity of IONIS-STAT3Rx | Approximately 28 Days after last dose of IONIS-STAT3Rx
  Measured by RECIST in the study population who have measurable disease or relevant disease specific response criteria
Pharmacokinetics-Cmax | Approximately 28 days after last dose of IONIS-STAT3Rx
  Maximum observed drug concentration (Cmax)
STAT3 and other biomarkers | Approximately 28 days after last dose of IONIS-STAT3Rx
  The effect of treatment with IONIS-STAT3Rx on phospho-STAT3 and other biomarkers
Pharmacokinetics - Tmax | Approximately 28 days after last dose of IONIS-STAT3Rx
  Time taken to reach Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Steve Hughes, MD, Study Director — Ionis Pharmaceuticals, Inc.
Locations (9):
- United States (9):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Yale Cancer Center, New Haven, Connecticut
  - Blood and Marrow Transplant Group of Georgia at Northside Hospital, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Reilley MJ, McCoon P, Cook C, Lyne P, Kurzrock R, Kim Y, Woessner R, Younes A, Nemunaitis J, Fowler N, Curran M, Liu Q, Zhou T, Schmidt J, Jo M, Lee SJ, Yamashita M, Hughes SG, Fayad L, Piha-Paul S, Nadella MVP, Xiao X, Hsu J, Revenko A, Monia BP, MacLeod AR, Hong DS. STAT3 antisense oligonucleotide AZD9150 in a subset of patients with heavily pretreated lymphoma: results of a phase 1b trial. J Immunother Cancer. 2018 Nov 16;6(1):119. doi: 10.1186/s40425-018-0436-5. PMID 30446007